CLINICAL TRIAL: NCT02130856
Title: An Integrated Toolkit to Save Newborn Lives in Pakistan
Brief Title: Newborn Kit to Save Lives in Pakistan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Grand Challenges Canada (Other); UBS Optimus Foundation (Other); Mother and Child Care Trust (MCCT), Pakistan (Unknown); Aga Khan University (Other); March of Dimes (Other)
Responsible Party: Principal Investigator, Shaun Morris, Associate Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1000042963
Record Dates: First submitted 2014-05-01; First posted 2014-05-05 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Neonatal Mortality
Keywords: Neonatal mortality; Neonatal kit; Pakistan; Randomized Control Trial; Chlorhexidine; ThermoSpot; Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neonatal Kit (Experimental): The neonatal kit will contain a clean birth kit to be used at the time of delivery either at home or in a facility, 4% chlorhexidine (CHX) lotion, sunflower oil emollient, ThermoSpot, a Mylar infant sleeve, and a reusable, non-electric, heating device. Lady Health Workers will be equipped with a hand held electric scale to identify low birth weight newborns.
  Interventions: Device: Neonatal kit
- Control (Standard care) (No Intervention): In the control arm, Lady Health Workers will visit the home according to the regular schedule (same as in the intervention clusters) and will deliver the standard post-natal care consisting of:
  1. be present at delivery (though not conduct the delivery) and thorough examination of newborn and mother post delivery
  2. check mother for vaginal bleeding and abnormal blood pressure and make referral to nearest health facility as appropriate
  3. refer any newborn with congenital anomaly or evidence of asphyxia
  4. if unable to attend delivery for any reason, visit within first 24 hours post delivery
  5. assess newborn in first month of life during visits and provide basic treatment for acute respiratory infections, pneumonia, and diarrhea in the home
  6. encourage breastfeeding

INTERVENTIONS:
Device: Neonatal kit — Contents of the neonatal kit:
  1. Clean birth kit: sterile blade, a clean plastic square, plastic gloves, hand soap, and cord ties/clamp.
  2. 4% Chlorhexidine (CHX) lotion (15 mL) and a bag of cotton balls.
  3. Sunflower oil emollient (50 mL)
  4. ThermoSpot
  5. Mylar infant sleeve
  6. Click to heat warmer (http://www.heatinaclick.ca/products/pocket_size.html) in a fitted cloth pouch.
  7. Handheld electric scale with suspended cloth sling. The scale will not be included with the kit but rather one will be issued to each Lady Health Worker.
  Arms: Neonatal Kit

SUMMARY:
There are over 3 million annual neonatal deaths. Approximately 2/3 of neonatal deaths are due to infection, low birth weight (LBW), and prematurity. Low tech but high impact interventions and commodities used in unconventional ways could save hundreds of thousands of newborn lives. We propose an integrated evidence-based toolkit usable by community health workers (CHW) to reduce neonatal deaths. The kit will include: Chlorhexidine to be applied to the umbilical stump, sunflower oil emollient to be applied to the skin, ThermoSpot to identify hypo/hyperthermia, and a Mylar infant sleeve with non-electric warmer.

DETAILED DESCRIPTION:
Over 3 million global neonatal deaths are reported annually. While significant progress has been made over the past decade towards reducing overall under 5 mortality, very little progress has been made towards the reduction of neonatal deaths, which represent about 40% of all deaths in children under the age of 5. The majority of neonatal deaths occur in rural areas of low-income countries and approximately two thirds are due to infection and complications relating to low birth weight (LBW) and prematurity.

In Pakistan, it is estimated that over 200,000 newborns die each year before they reach the end of their first month of life, representing nearly 58% of all deaths among children under the age of five. The risk of neonatal death in Pakistan is higher in rural areas than in urban areas; the neonatal mortality rate (NMR) in rural areas is 55 per 1,000 live births compared to 48 per 1,000 live births in urban areas. NMR in Pakistan is also associated with poverty; the NMR in highest wealth quintile is 38 compared to 63 per 1000 live births in lowest wealth quintile.

In resource poor settings, newborns are most often delivered at home and receive minimal specific medical care, measurement, or monitoring. In these areas, geography, infrastructure, and poverty often effectively prevent access to health centers and care. Home outreach with trained Community health workers (CHWs) is increasingly recognized as the mainstay for provision of maternal and newborn care in these settings. Many proven, cost-effective ways to save the lives of newborns exist, however, they are not always available to those who need them most nor have they been packaged into a single portable kit that can be easily used in the home-setting. Such a portable kit consisting of low cost, evidence-based interventions for use in the home has tremendous potential to improve health status and decrease NMR.

In this study, the investigators hypothesize that the implementation of an integrated evidence-based toolkit by CHWs will reduce neonatal deaths by at least 40% through a reduction in both infectious causes of death and those associated with prematurity and LBW. Furthermore, the investigators propose that there will be an additive effect from the mortality benefit of specific kit components. The portable kit will contain a clean birth kit to be used at the time of delivery either at home or in a facility, 4% chlorhexidine (CHX) lotion, sunflower oil emollient, ThermoSpot, a Mylar infant sleeve, and a reusable, non-electric, heating device. CHWs will be equipped with a hand held electric scale to identify LBW newborns.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women in parts of study clusters covered by Lady Health Worker program and their home- or facility-born live newborns
* Mother intending to maintain residence in study area for first month of newborn's life

Exclusion Criteria:

* Failure to provide consent to enroll in study (intervention or control clusters)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8518 (Actual)
Dates: Start 2014-04; Primary Completion 2017-02-26 (Actual); Study Completion 2017-02-26 (Actual)

PRIMARY OUTCOMES:
Neonatal mortality | During phase I of the study: Day 1 (or as soon as possible after notification of birth), 3, 7, 14, and 28 of life. During phase II of the study: Day 8 and day 28 of life.
  Death from any cause within the first 28 days of life

SECONDARY OUTCOMES:
Incidence of omphalitis | During phase I of the study: Day 1 (or as soon as possible after notification of birth), 3, 7, 14, and 28 of life. During phase II of the study: Day 8 and day 28 of life.
  Incidence of omphalitis where omphalitis is defined as:
  1. None (no redness or swelling)
  2. Mild (inflammation limited to the cord stump)
  3. Moderate (inflammation extending less than 2cm to the skin at the base of the cord stump)
  4. Severe (inflammation extending more than 2cm from the cord stump)
Incidence of severe infection | During phase I of the study: Day 1 (or as soon as possible after notification of birth), 3, 7, 14, and 28 of life. During phase II of the study: Day 8 and day 28 of life.
  Incidence of severe infection is defined as:
  a) Convulsions OR fast breathing (60 breaths per minute or more) OR severe chest indrawing OR movement only when stimulated or no movement at all OR not feeding at all for at least 12 hours.
Cases of hypothermia identified | During phase I of the study: Day 1 (or as soon as possible after notification of birth), 3, 7, 14, and 28 of life. During phase II of the study: Day 8 and day 28 of life.
  Hypothermia defined using ThermoSpot as:
  1. Moderate hypothermia: pale green and red face (35C to 36C)
  2. Severe hypothermia: black face (<35C)
Cases of hyperthermia identified | During phase I of the study: Day 1 (or as soon as possible after notification of birth), 3, 7, 14, and 28 of life. During phase II of the study: Day 8 and day 28 of life.
  Hyperthermia defined using ThermoSpot as:
  a) Hyperthermia: blue face (>39C)
Number of low birth weight (LBW) newborns identified | During phase I of the study: Day 1 (or as soon as possible after notification of birth), 3, 7, 14, and 28 of life. During phase II of the study: Day 8 and day 28 of life.
  LBW is defined as:
  <2500 grams at first weighing
Health Facility Use | During phase I of the study: Day 1 (or as soon as possible after notification of birth), 3, 7, 14, and 28 of life. During phase II of the study: Day 8 and day 28 of life.
Neurodevelopmental score at 12 months of age | Month 12 of life (only during phase I of the study)
  Assessed by the Bayley Scale of Infant Development III (BSID III).

CONTACTS AND LOCATIONS:
Overall Officials: Shaun K. Morris, MD, MPH, Principal Investigator — The Hospital for Sick Children, Toronto; Zulfiqar A. Bhutta, PhD, MBBS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Pakistan

REFERENCES:
- [Background] Liu L, Johnson HL, Cousens S, Perin J, Scott S, Lawn JE, Rudan I, Campbell H, Cibulskis R, Li M, Mathers C, Black RE; Child Health Epidemiology Reference Group of WHO and UNICEF. Global, regional, and national causes of child mortality: an updated systematic analysis for 2010 with time trends since 2000. Lancet. 2012 Jun 9;379(9832):2151-61. doi: 10.1016/S0140-6736(12)60560-1. Epub 2012 May 11. PMID 22579125
- [Background] Khan A, Kinney MV, Hazir T, Hafeez A, Wall SN, Ali N, Lawn JE, Badar A, Khan AA, Uzma Q, Bhutta ZA; Pakistan Newborn Change and Future Analysis Group. Newborn survival in Pakistan: a decade of change and future implications. Health Policy Plan. 2012 Jul;27 Suppl 3:iii72-87. doi: 10.1093/heapol/czs047. PMID 22692418
- [Background] Bhutta ZA, Rehman S. Perinatal care in Pakistan: a situational analysis. J Perinatol. 1997 Jan-Feb;17(1):54-9. PMID 9069067
- [Background] Mullany LC, Darmstadt GL, Khatry SK, Katz J, LeClerq SC, Shrestha S, Adhikari R, Tielsch JM. Topical applications of chlorhexidine to the umbilical cord for prevention of omphalitis and neonatal mortality in southern Nepal: a community-based, cluster-randomised trial. Lancet. 2006 Mar 18;367(9514):910-8. doi: 10.1016/S0140-6736(06)68381-5. PMID 16546539
- [Background] Soofi S, Cousens S, Imdad A, Bhutto N, Ali N, Bhutta ZA. Topical application of chlorhexidine to neonatal umbilical cords for prevention of omphalitis and neonatal mortality in a rural district of Pakistan: a community-based, cluster-randomised trial. Lancet. 2012 Mar 17;379(9820):1029-36. doi: 10.1016/S0140-6736(11)61877-1. Epub 2012 Feb 8. PMID 22322126
- [Background] Arifeen SE, Mullany LC, Shah R, Mannan I, Rahman SM, Talukder MR, Begum N, Al-Kabir A, Darmstadt GL, Santosham M, Black RE, Baqui AH. The effect of cord cleansing with chlorhexidine on neonatal mortality in rural Bangladesh: a community-based, cluster-randomised trial. Lancet. 2012 Mar 17;379(9820):1022-8. doi: 10.1016/S0140-6736(11)61848-5. Epub 2012 Feb 8. PMID 22322124
- [Background] Darmstadt GL, Saha SK, Ahmed AS, Ahmed S, Chowdhury MA, Law PA, Rosenberg RE, Black RE, Santosham M. Effect of skin barrier therapy on neonatal mortality rates in preterm infants in Bangladesh: a randomized, controlled, clinical trial. Pediatrics. 2008 Mar;121(3):522-9. doi: 10.1542/peds.2007-0213. PMID 18310201
- [Background] Green DA, Kumar A, Khanna R. Neonatal hypothermia detection by ThermoSpot in Indian urban slum dwellings. Arch Dis Child Fetal Neonatal Ed. 2006 Mar;91(2):F96-8. doi: 10.1136/adc.2005.078410. Epub 2005 Sep 13. PMID 16159955
- [Background] Krautheim AB, Jermann TH, Bircher AJ. Chlorhexidine anaphylaxis: case report and review of the literature. Contact Dermatitis. 2004 Mar;50(3):113-6. doi: 10.1111/j.0105-1873.2004.00308.x. PMID 15153122
- [Background] Rosenberg A, Alatary SD, Peterson AF. Safety and efficacy of the antiseptic chlorhexidine gluconate. Surg Gynecol Obstet. 1976 Nov;143(5):789-92. PMID 982260
- [Background] Garland JS, Alex CP, Mueller CD, Otten D, Shivpuri C, Harris MC, Naples M, Pellegrini J, Buck RK, McAuliffe TL, Goldmann DA, Maki DG. A randomized trial comparing povidone-iodine to a chlorhexidine gluconate-impregnated dressing for prevention of central venous catheter infections in neonates. Pediatrics. 2001 Jun;107(6):1431-6. doi: 10.1542/peds.107.6.1431. PMID 11389271
- [Background] Darmstadt GL, Mao-Qiang M, Chi E, Saha SK, Ziboh VA, Black RE, Santosham M, Elias PM. Impact of topical oils on the skin barrier: possible implications for neonatal health in developing countries. Acta Paediatr. 2002;91(5):546-54. doi: 10.1080/080352502753711678. PMID 12113324
- [Background] Darmstadt GL, Saha SK, Ahmed AS, Chowdhury MA, Law PA, Ahmed S, Alam MA, Black RE, Santosham M. Effect of topical treatment with skin barrier-enhancing emollients on nosocomial infections in preterm infants in Bangladesh: a randomised controlled trial. Lancet. 2005 Mar 19-25;365(9464):1039-45. doi: 10.1016/S0140-6736(05)71140-5. PMID 15781099
- [Background] Lawn JE, Kinney MV, Black RE, Pitt C, Cousens S, Kerber K, Corbett E, Moran AC, Morrissey CS, Oestergaard MZ. Newborn survival: a multi-country analysis of a decade of change. Health Policy Plan. 2012 Jul;27 Suppl 3:iii6-28. doi: 10.1093/heapol/czs053. PMID 22692417
- [Derived] Duby J, Pell LG, Ariff S, Khan A, Bhutta A, Farrar DS, Bassani DG, Hussain M, Bhutta ZA, Soofi S, Morris SK. Effect of an integrated neonatal care kit on cause-specific neonatal mortality in rural Pakistan. Glob Health Action. 2020 Dec 31;13(1):1802952. doi: 10.1080/16549716.2020.1802952. PMID 32838701
- [Derived] Turab A, Pell LG, Bassani DG, Soofi S, Ariff S, Bhutta ZA, Morris SK. The community-based delivery of an innovative neonatal kit to save newborn lives in rural Pakistan: design of a cluster randomized trial. BMC Pregnancy Childbirth. 2014 Sep 8;14:315. doi: 10.1186/1471-2393-14-315. PMID 25201572